CLINICAL TRIAL: NCT02368041
Title: Utility of Thenar Near Infrared Spectroscopy (NIRS) in Pediatric Patients With Heart Failure
Status: Recruiting | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB202200657; IRB201400800 (Other: UF IRB-01)
Record Dates: First submitted 2015-02-13; First posted 2015-02-20 (Estimated); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- InSpectraTM StO2: InSpectraTM StO2 monitor manufactured by Hutchinson Technology Inc. to measure the baseline StO2 level after applying the noninvasive probe to the thenar eminence. After a stable reading is obtained a blood pressure cuff will be inflated 40 mmHg above the obtained systolic pressure and the rate of desaturation (Rdes; % × sec-1) will be recorded. After 3 minutes or once the StO2 level comes to zero, whichever is earlier the cuff pressure will be released instantaneously and the rate of reperfusion (Rres; % × sec-1) will be measured. The measurement will be continued until the StO2 returns to the baseline value.
  Interventions: Device: InSpectraTM StO2 monitor

INTERVENTIONS:
Device: InSpectraTM StO2 monitor — InSpectraTM StO2 monitor manufactured by Hutchinson Technology Inc. to measure the baseline StO2 level after applying the noninvasive probe to the thenar eminence. After a stable reading is obtained a blood pressure cuff will be inflated 40 mmHg above the obtained systolic pressure and the rate of desaturation (Rdes; % × sec-1) will be recorded. After 3 minutes or once the StO2 level comes to zero, whichever is earlier the cuff pressure will be released instantaneously and the rate of reperfusion (Rres; % × sec-1) will be measured. The measurement will be continued until the StO2 returns to the baseline value.

SUMMARY:
This is a single-center, non-randomized study.The study staff will use the InSpectraTM tissue oxygen saturation (StO2) monitor manufactured by Hutchinson Technology to measure baseline StO2 levels after applying the noninvasive probe to the thenar eminence. After a stable reading is obtained, a blood pressure cuff will be inflated 40 mmHg above the obtained systolic pressure and the rate of desaturation (Rdes; % × sec-1) will be recorded. After 3 minutes or once the StO2 level comes to zero (whichever is earlier), the cuff pressure will be released and the rate of reperfusion (Rres; % × sec-1) will be measured. The investigators hypothesize that heart failure in children causes a baseline lower thenar tissue oxygen saturation (StO2), a faster rate of desaturation (Rdes) and a prolonged rate of reperfusion (Rres). The investigators also hypothesize that these changes will correlate with the severity of heart failure. The results of this study will provide groundwork for studies looking at correlation of therapy modification based on the combination thenar StO2 and clinical presentation.

DETAILED DESCRIPTION:
Heart failure patients seen in the Pediatric Cardiology Congenital Heart Center will be enrolled into the study after obtaining informed consent on the day of their evaluation. The primary pediatric cardiologist following the patient will evaluate the need for regular investigations like blood work, electrocardiogram and echocardiogram. The study staff will use the InSpectraTM tissue oxygen saturation (StO2) monitor manufactured by Hutchinson Technology to measure the baseline StO2 level after applying the noninvasive probe to the thenar eminence. After a stable reading is obtained a blood pressure cuff will be inflated 40 mmHg above the obtained systolic pressure and the rate of desaturation (Rdes; % × sec-1) will be recorded. After 3 minutes or once the StO2 level comes to zero (whichever is earlier), the cuff pressure will be released and the rate of reperfusion (Rres; % × sec-1) will be measured. Similar measurements will be obtained from an otherwise healthy cohort of children who present to the Pediatric Cardiology Congenital Heart Center for evaluation of a heart murmur or chest pain. The patient's treating physician and care providers will be blinded to the study test results. All clinical care will be at the discretion of the patient's treating physicians. Only StO2 levels will be obtained using the non-invasive probe placed on the thenar eminence for the purpose of the study.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure patients under 25 years of age with a diagnosis of cardiomyopathy, myocarditis or univentricular palliation for congenital heart disease who are stable on their medical management will be enrolled.

Exclusion Criteria:

1. Patients presenting with acute deterioration in clinical status
2. Patients with active infection
3. Patients with autoimmune vasculitis disorder
4. Patients with limb deformities and painful disorders of extremities
5. Patients with underlying bone disorders, (e.g. osteogenesis imperfecta)
6. Patients with severe anemia (Hb <7g/dL)
7. Patients with peripheral vascular disease which can alter the microcirculation

Max Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Stable Heart failure patients under 25 years of age with a diagnosis of cardiomyopathy, myocarditis or univentricular palliation for congenital heart disease in a primary pediatric cardiologist office
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2015-05 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2026-05-10 (Estimated)

PRIMARY OUTCOMES:
Baseline StO2 percentage | Day 1
  The study staff will use the InSpectraTM StO2 monitor manufactured by Hutchinson Technology to measure the baseline StO2 level after applying the noninvasive probe to the thenar eminence

SECONDARY OUTCOMES:
Occlusion- rate of desaturation (Rdes) of StO2 levels | Day 1
  After a stable baseline reading is obtained a blood pressure cuff will be inflated 40 mmHg above the obtained systolic pressure and the rate of desaturation (Rdes; % × sec-1) will be recorded for 3 min or until the StO2 level comes to zero (whichever is earlier).
Recovery- rate of reperfusion (Rres) of StO2 levels | Day 1
  After 3 minutes from occlusion or once the StO2 level comes to zero (whichever is earlier), the cuff pressure will be released and the rate of reperfusion (Rres; % × sec-1) will be measured for approximately 3 min.

CONTACTS AND LOCATIONS:
Overall Officials: Dipankar Gupta, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant will not be shared to avoid risk of loss of confidentiality.